CLINICAL TRIAL: NCT00165308
Title: A Feasibility Study of Tamoxifen Prevention of Breast Cancer in Hodgkin's Disease Survivors
Brief Title: Tamoxifen in the Prevention of Breast Cancer in Hodgkin's Disease Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Judy E. Garber, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00-253
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Hodgkin's Disease; Breast Cancer
Keywords: Hodgkin's disease; breast cancer prevention; tamoxifen
MeSH Terms: conditions — Hodgkin Disease; Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tamoxifen (Experimental): Single arm: Tamoxifen 20mg daily
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Given orally, daily for one year.

SUMMARY:
The purpose of this study is determine whether or not tamoxifen reduces the chance of Hodgkin's Disease survivors developing breast cancer.

DETAILED DESCRIPTION:
* Patients will receive tamoxifen orally once daily to be taken at home for 1 year. They will be asked to complete a daily drug log to keep track of the pills taken or missed.
* Patients will also be asked to give a blood/DNA sample which will be stored for possible further testing for the presence of cancer related genes that are known nor or discovered in the future.
* Patients will also receive a mammogram that will be reviewed by study officials.
* Side effects will be monitored every 2 months for one year, between visits to the clinic.
* A follow-up visit will be conducted at the 6 month mark and includes a physical exam, blood work, health and wellness surveys)
* A follow-up visit will be performed at the 1 year mark and includes a mammogram, gynecological exam, physical exam, blood work, health and wellness surveys.
* Patients active participation will be for 1 year. However, tamoxifen has been shown to be effective after a 5-year course in other women at increased risk for breast cancer, the patient may decide to stay on tamoxifen for 4 additional years.

ELIGIBILITY:
Inclusion Criteria:

* Females diagnosed with Hodgkin's Disease at age < 35 years
* > 5 years from mantle or chest radiation
* Current age > 30 years
* Has completed childbearing
* Willingness to discontinue use of oral contraceptives or other hormonal contraception for duration of the study

Exclusion Criteria:

* History of secondary malignancy after Hodgkin's disease, except thyroid cancer of basal cell cancer
* Recurrence of Hodgkin's disease in the 5 years before study entry
* Current participation in any other cancer prevention study
* Current or prior use of tamoxifen
* Current use of coumadin
* History of deep venous thrombosis, pulmonary embolism, or a condition known to be associated with hypercoagulability
* History of cerebrovascular accident
* History of macular degeneration
* Current use of chemotherapy for benign disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2001-04; Primary Completion 2004-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of a randomized trial testing the effectiveness of tamoxifen in reducing the risk of radiogenic breast cancer. | 2 years

SECONDARY OUTCOMES:
To determine the safety and effect on quality of life in participating women. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Judy Garber, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute; Lisa Diller, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Boucher AA, Blaes AH. Prophylactic mastectomy: a treatment alternative for Hodgkin survivors? Clin Breast Cancer. 2013 Oct;13(5):307-8. doi: 10.1016/j.clbc.2013.06.001. Epub 2013 Jul 26. No abstract available. PMID 23891588